CLINICAL TRIAL: NCT06190548
Title: Clinical Outcomes of Hypervirulent Carbapenem-resistant Klebsiella Pneumoniae Infection: a Single-centre Cohort Study With Multiplex Analyses in China
Brief Title: Clinical Outcomes of Hypervirulent Carbapenem-resistant Klebsiella Pneumoniae Infection
Acronym: HVCRKP
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ya Hu, Dr., West China Hospital
Other Study IDs: SichuanU; 81861138055 (Other: National Natural Science Foundation of China)
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Infection, Bacterial
Keywords: Klebsiella pneumoniae; hypervirulent; clinical outcome
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Clinical samples which were identified as containing CRKP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cCRKP: Patients with classic CRKP infection
- hvCRKP: Patients with hypervirulent CRKP infection

SUMMARY:
The goal of this observational study is to learn about the risk factors of mortality for CRKP infected patients, and to compare the clinical outcomes between hvCRKP infection and cCRKP infection. The main question it aims to answer is • Whether hypervirulence would add value to cCRKP infection and cause worse outcomes? Participants data will be collected through medical records.

DETAILED DESCRIPTION:
We conducted an observational cohort study comprising three-year (2019-2022) data in a Chinese university hospital. We performed genome sequencing for CRKP strains, compared adult patients infected by hvCRKP with those by non-hypervirulent "classical" CRKP (cCRKP), and used propensity score matching (PSM) for imbalanced baseline characteristics. We defined 30-day all-cause and attributed mortalities and 30-day ranking outcomes (death, no response/progress, remission) as primary outcomes and post-infection stay and survival as secondary outcomes. We constructed mortality-predicting models and performed subgroup analyses for CRKP of the dominant sequence or capsular type or with varied virulence profiles and for patients with bloodstream or lower respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18-year-old) with CRKP infections were included.

Exclusion Criteria:

* younger than 18 years old; clinical samples were identified to contain CRKP but were sentenced to be colonization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CRKP infection
Sampling Method: Non-Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  The mortality of patients 30-days after CRKP infection
The number of participants with status | 30 days
  The status of patients 30 days after CRKP infection, including death, no response or progress, and remission.

SECONDARY OUTCOMES:
length of stay (LOS) in the hospital | 30 days
  length of stay of the patients
post-infection survival | 30 days
  Survival of patients after CRKP infection

CONTACTS AND LOCATIONS:
Overall Officials: Center of infectious diseases, Study Director — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
The original data might be shared in the form of an article attachment, but it was not decided for now.